CLINICAL TRIAL: NCT04814160
Title: Ridge Splitting and Simultaneous Implant Placement With Autogenous Bone and Bioactive Glass for the Treatment of Maxillary Horizontal Bone Defects: A Randomised Clinical Trial
Brief Title: Autobone and Bioactive Glass With Ridge Splitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, lecturer of oral medicine and periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSBG2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Horizontal Alveolar Ridge Deficiency
Keywords: Ridge split; dental implant; piezosurgery; bioactive glass; autogenous bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous bone graft (Active Comparator): autogenous bone graft for augmenting bone defects around dental implants placed simultaneously with ridge splitting
  Interventions: Procedure: autogenous bone graft
- mix of bioactive glass and autogenous bone graft (Experimental): 1:1 mix of bioactive glass and autogenous bone graft for augmenting bone defects around dental implants placed simultaneously with ridge splitting
  Interventions: Procedure: mixture of bioactive glass and autogenous bone graft

INTERVENTIONS:
Procedure: mixture of bioactive glass and autogenous bone graft — bone expansion was performed and autogenous bone mixed with bioactive glass was used to augment the intercortical bone defect after ridge splitting and simultaneous dental implants
  Arms: mix of bioactive glass and autogenous bone graft
Procedure: autogenous bone graft — bone expansion was performed and autogenous bone alone was used to augment the intercortical bone defect after ridge splitting and simultaneous dental implants
  Arms: autogenous bone graft

SUMMARY:
Objective: To compare the use of autogenous bone graft versus autogenous bone graft mixed with bioactive glass bone graft in the treatment of maxillary anterior horizontal bone defects by ridge splitting technique combined with simultaneous implant placement.

Materials and methods: Twenty-two patients were divided randomly into two groups; control group and study group. In control group, bone expansion was performed and autogenous bone was used to augment the intercortical bone defect. In study group, bone expansion was performed and autogenous bone mixed with bioactive glass was used to augment the intercortical bone defect. In both groups, the implants were inserted simultaneously with ridge splitting. 6 months after implant placement, the mean bone width and alveolar bone loss values were evaluated. Statistical analysis using paired Student's t- test to compare results within the same group of patients, whereas, independent samples t-test was used to compare variables between the two groups

DETAILED DESCRIPTION:
Participants' selection:

22 patients, aged from 18 to 50 years, were selected in this prospective, randomized and blinded clinical trial from the Outpatient Clinic of the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Kafrelsheikh University. Those subjects had inadequate bone volume for implant placement due to width insufficiency of maxillary anterior alveolar ridges. The research ethical committee of Faculty of Dentistry, Kafrelsheikh University approved the study (KD/06/21). Research procedures were explained to all patients, and they agreed to participate in the study and signed the appropriate informed consent form. The inclusion criteria implemented for patient selection were good general health at the time of surgery; at least 3months postextraction healing period; and horizontally compromised maxillary anterior alveolar ridges (at least 3mm bone width and 13mm bone height). The criteria of patients exclusion were vertical bone defect; thick labial cortex with less cancellous bone inside; obvious undercut on the labial/buccal side; uncontrolled periodontal conditions; history of radiotherapy in the head and neck region; uncontrolled diabetes mellitus or other systematic disorders; smokers; pregnancy; non-compliant patients; and allergic reaction to the used medications.

Pre-surgical therapy and grouping Pre-surgical therapy consisted of a thorough full-mouth scaling and root planning. Patients were randomly assigned immediately before surgery into two groups (11 patients each) by computer-assessed randomization software (Random Allocation Software, Version 1.0). Control group received ridge splitting with simultaneous implant placement in combination with autogenous bone graft alone, while study group used (1:1) mixture of autogenous and bioactive glass bone grafts. Bone volume was assessed two weeks before operation using CBCT (Scanora 3D, Soredex Oy, Tuusula, Finland).

Surgical procedure:

Operations were performed under local anesthesia. Mid-crestal incision followed by full thickness flap reflection to expose surgical site. Mid crestal cut using piezo-surgery unit (Piezotome® Cube, ACTEON®, Acteon Group Ltd, Norwich, England). Then, the cut was extended deep to the length of implant. Then, ridge was expanded progressively using bone wedges (Microdent Implant System, Spain). Implant location was marked, with a buccal bony wall as uniformly thick (>1 mm) as possible to avoid bone fracture. The implant site was prepared and 3.75*13 mm dental implant fixture (Humana Dental Implants & Accessories GmbH, Germany) was placed stably in between the two bony plates.

Autogenous bone harvesting:

Incision was made at mucogingival junction in the symphysis area followed by full thickness flap reflection, and then corticocancellous bone was harvested using a trephine drill. Finally the flap was sutured by interrupted and horizontal mattress suture by 3-0 black silk.

In control group, harvested autogenous bone graft was used for augmentation of the gap between buccal and lingual plates. Study group received the same way of treatment except using (1:1) mixture of the harvested autogenous bone with bioactive glass bone graft (BonyGlass, Pharma-Excellence, Egypt). The wound was completely closed in a tension-free way. All surgeries were performed by the same operator.

Postoperative care:

Patients were prescribed amoxicillin-clavulanic acid 1g. every 12hours antibiotic (Augmentin 1g, SmithKline Beecham Pharmaceuticals), and 0.12% chlorhexidine hydrochloride mouth wash twice daily (Hexitol, ADCO, Cairo, A.R.E). The sutures were removed 14days postoperatively. No removable denture was allowed to wear for 2weeks.

6months postoperatively, clinical evaluation was recorded including implant survival, presence of infection, pain, tenderness or wound dehiscence. CBCT was taken at 6months postoperatively to evaluate ridge width and bone level. All clinical and radiographic measurements were recorded by one calibrated masked examiner.

Study variables The primary outcome variable was linear changes in the marginal bone surrounding the implants and alveolar ridge width, taken from cross-sectional and longitudinal CBCT images. Bone heights and width were assessed preoperatively and after 6months postoperatively using the CBCT images.

Statistical analysis:

Sample size calculation was undertaken via G power version 3.1 statistical software based on the following pre-established parameters: an alpha-type error of 0.05, a power test of 0.80, a total sample of 22 subjects (11 subjects for each group) appeared to be sufficient.

The statistical analysis was performed using IBM SPSS version 20 software (IBM Corp., Armonk, NY, USA). Data were presented as the mean+stanstandard deviation. The paired Student's t- test was used to compare the obtained results within the same group of patients at 2 different intervals. The independent samples t-test was used to compare variables between the two groups. In all tests, the result was considered statistically significant if the P-value was <0.05.

ELIGIBILITY:
Inclusion Criteria:

* good general health at the time of surgery
* at least 3months postextraction healing period
* horizontally compromised maxillary anterior alveolar ridges (at least 3mm bone width and 13mm bone vertical height).

Exclusion Criteria:

* vertical bone defect
* thick labial cortex with less cancellous bone inside
* obvious undercut on the labial/buccal side
* uncontrolled periodontal conditions
* history of radiotherapy in the head and neck region
* uncontrolled diabetes mellitus or other systematic disorders
* smokers
* pregnancy
* non-compliant patients
* allergic reaction to the used medications.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical measurements of pain intensity | 6 months
  pain intensity verbal rating scale either mild, moderate or sever
Clinical incidence of implants mobility | 6 months
  Implants mobility
measuring the survival rates | 6 months
  survival rates of implants

SECONDARY OUTCOMES:
radiographic results of bone width and height | 6 months
  evaluation of bone width and height using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Egypt

REFERENCES:
- [Derived] Elamrousy W, Osama M, Issa DR. Autogenous Bone and Bioactive Glass around Implants Placed Simultaneously with Ridge Splitting for the Treatment of Horizontal Bony Defects: A Randomised Clinical Trial. Int J Dent. 2021 Jul 28;2021:2457328. doi: 10.1155/2021/2457328. eCollection 2021. PMID 34367287